CLINICAL TRIAL: NCT03359486
Title: Pilot Feasibility Study of Focused Psychosocial Support to Improve the Psychosocial Well-being and Functioning of Adults Affected by Humanitarian Crisis in Nepal
Brief Title: Pilot Feasibility Study of Psychosocial Support to Improve Well-being of Adults in Humanitarian Crises in Nepal
Acronym: PM+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: World Health Organization (Other); Transcultural Psychosocial Organization Nepal (Other); Duke University (Other); King's College London (Other)
Responsible Party: Principal Investigator, Brandon Kohrt, Associate Professor of Psychiatry, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERC.0002817
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group problem management plus (Experimental): Five sessions of group low intensity psychological intervention
  Interventions: Behavioral: Group problem management plus
- Enhanced treatment as usual (Active Comparator): Referral to primary health care workers trained in mental health Gap Action Programme.
  Interventions: Behavioral: Group problem management plus; Behavioral: Enhanced treatment as usual

INTERVENTIONS:
Behavioral: Group problem management plus — Low intensity group psychological intervention including stress management, behavioral activation, problem solving, and strengthening social support
Behavioral: Enhanced treatment as usual — Referral to primary care workers trained in mental health Gap Action Program Implementation Guide
  Other Names: mental health Gap Action Program-Implementation Guide
  Arms: Enhanced treatment as usual

SUMMARY:
This is a pilot feasibility study of group problem management plus, a low-intensity psychological intervention, delivered in five sessions to adults affected by humanitarian crises. The current study will evaluate feasibility and acceptability of the intervention to determine procedures and content for a subsequent full trial using a cluster-randomized design of group problem management plus versus enhanced treatment as usual.

DETAILED DESCRIPTION:
Counselling programmes used in many humanitarian settings are often non-specific with unknown efficacy and safety. Only a few interventions in humanitarian crises have been rigorously tested, and most studied interventions focused on posttraumatic stress disorder. Beyond posttraumatic stress disorder, individuals may have a range of problems including depression, anxiety, and not being able to do daily tasks necessary for survival and recovery. However, interventions are often limited since they tend to target only a single outcome, are usually of longer duration (8-16 sessions) or require professionals.

In low resourced settings interventions need to be short of duration, and be carried out by lay people in the communities to make them sustainable and feasible to implement on a broader scale. World Health Organization aims to develop a range of low-intensity scale-able psychological interventions that address these issues, as part of its mental health Gap Action Program. As a first step a simplified psychological intervention Problem Management Plus (PM+) has been developed. It has 4 core features that make the intervention suitable for low resourced setting exposed to adversities. First, it is brief intervention (5-sessions), delivered individually or in groups; second, it can be delivered by paraprofessionals (high school graduates with no mental health experience), using the principle of task shifting/ task sharing; third, it is designed as a trans-diagnostic intervention, addressing a range of client identified emotional (e.g. depression, anxiety, traumatic stress, general stress) and practical problems; fourth, it is designed for people in low-income country communities affected by any kind of adversity (e.g. violence, disasters), not just focusing on a single kind of adversity.

Recent PM+ trails in Pakistan and Kenya have indicated PM+ to be effective in diminishing depression and anxiety and improving people's functioning and self-selected, culturally relevant outcomes. In this project Group PM+ will be piloted in a district in Nepal, which was affected by the 2015 earthquakes in Nepal. The current pilot study will evaluate the acceptability and feasibility of Group PM+ in Nepal to informant a subsequent pragmatic cluster randomized controlled trial. This exploratory cluster randomized controlled trial (cluster randomized controlled trial) will be conducted to gather information about the feasibility, safety and delivery of the intervention in the Nepali community settings; and to identify issues around training, supervision and outcomes measures. This research strategy is informed by the United Kingdom Medical Research Council framework for the development of complex interventions, which recognizes iterations of: a) Intervention Development; b) Feasibility and Piloting; c) Evaluation; and d) Implementation. This framework recommends to first conduct feasibility and randomized pilot studies before conducting large scale trials. In this way possible problems of acceptability, compliance, delivery of the intervention, recruitment and retention can be detected before the large definitive scale trail is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. score >2 on General Health Questionnaire (dichotomous item scoring method)
2. score >16 on World Health Organization Disability Assessment Scale

Exclusion Criteria:

1. Presence of a severe mental disorder (e.g., psychosis)
2. Alcohol use disorder (score >16 on the alcohol use disorders identification test (AUDIT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported gender
Enrollment: 120 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Depression - Patient Health Questionnaire | 1 week post-intervention
  9-item measure of depression symptoms, culturally and clinically validated in Nepal

SECONDARY OUTCOMES:
Daily functioning - World Health Organization Disability Assessment Scale | 1 week post-intervention
  12-item assessment ability to engage in daily activities, previously used in numerous studies in Nepal
General psychological distress - General Health Questionnaire | 1 week post-intervention
  12-item measure of general psychological distress, previously validated for use in Nepal
Posttraumatic Stress Disorder - Posttraumatic Stress Disorder Checklist | 1 week post-intervention
  8-tem measure of post-traumatic stress symptoms validated for use in Nepal
Personalized Measure of Distress - Psychological Outcome Profiles | 1 week post-intervention
  3-item measure of personalized distress and problems, 4-items post-treatment
Culture-specific general psychological distress - Nepali Psychosocial and Mental Health Problems | 1 week post-intervention
  5-item measure of somatic symptoms of psychosocial and mental health problems validated in Nepal
Reducing Tension Checklist for Problem Management Plus Skills | 1 week post-intervention
  12-item measure of behavioral and psychosocial skills related to coping mechanisms

CONTACTS AND LOCATIONS:
Overall Officials: Mark van Ommeren, PhD, Study Director — World Health Organization
Locations (1):
- Transcultural Psychosocial Organization (TPO) Nepal, Kamalamai, Sindhuli, Nepal

IPD SHARING:
Plan to Share IPD: No
This will be shared for full trial.

REFERENCES:
- [Background] Bryant RA, Schafer A, Dawson KS, Anjuri D, Mulili C, Ndogoni L, Koyiet P, Sijbrandij M, Ulate J, Harper Shehadeh M, Hadzi-Pavlovic D, van Ommeren M. Effectiveness of a brief behavioural intervention on psychological distress among women with a history of gender-based violence in urban Kenya: A randomised clinical trial. PLoS Med. 2017 Aug 15;14(8):e1002371. doi: 10.1371/journal.pmed.1002371. eCollection 2017 Aug. PMID 28809935
- [Background] Khan MN, Hamdani SU, Chiumento A, Dawson K, Bryant RA, Sijbrandij M, Nazir H, Akhtar P, Masood A, Wang D, Wang E, Uddin I, van Ommeren M, Rahman A. Evaluating feasibility and acceptability of a group WHO trans-diagnostic intervention for women with common mental disorders in rural Pakistan: a cluster randomised controlled feasibility trial. Epidemiol Psychiatr Sci. 2019 Feb;28(1):77-87. doi: 10.1017/S2045796017000336. Epub 2017 Jul 10. PMID 28689511
- [Background] Hamdani SU, Ahmed Z, Sijbrandij M, Nazir H, Masood A, Akhtar P, Amin H, Bryant RA, Dawson K, van Ommeren M, Rahman A, Minhas FA. Problem Management Plus (PM+) in the management of common mental disorders in a specialized mental healthcare facility in Pakistan; study protocol for a randomized controlled trial. Int J Ment Health Syst. 2017 Jun 8;11:40. doi: 10.1186/s13033-017-0147-1. eCollection 2017. PMID 28603552
- [Background] Chiumento A, Hamdani SU, Khan MN, Dawson K, Bryant RA, Sijbrandij M, Nazir H, Akhtar P, Masood A, Wang D, van Ommeren M, Rahman A. Evaluating effectiveness and cost-effectiveness of a group psychological intervention using cognitive behavioural strategies for women with common mental disorders in conflict-affected rural Pakistan: study protocol for a randomised controlled trial. Trials. 2017 Apr 26;18(1):190. doi: 10.1186/s13063-017-1905-8. PMID 28441974
- [Background] Dawson KS, Schafer A, Anjuri D, Ndogoni L, Musyoki C, Sijbrandij M, van Ommeren M, Bryant RA. Feasibility trial of a scalable psychological intervention for women affected by urban adversity and gender-based violence in Nairobi. BMC Psychiatry. 2016 Nov 18;16(1):410. doi: 10.1186/s12888-016-1117-x. PMID 27863515
- [Background] Rahman A, Riaz N, Dawson KS, Usman Hamdani S, Chiumento A, Sijbrandij M, Minhas F, Bryant RA, Saeed K, van Ommeren M, Farooq S. Problem Management Plus (PM+): pilot trial of a WHO transdiagnostic psychological intervention in conflict-affected Pakistan. World Psychiatry. 2016 Jun;15(2):182-3. doi: 10.1002/wps.20312. No abstract available. PMID 27265713
- [Background] Sijbrandij M, Bryant RA, Schafer A, Dawson KS, Anjuri D, Ndogoni L, Ulate J, Hamdani SU, van Ommeren M. Problem Management Plus (PM+) in the treatment of common mental disorders in women affected by gender-based violence and urban adversity in Kenya; study protocol for a randomized controlled trial. Int J Ment Health Syst. 2016 May 31;10:44. doi: 10.1186/s13033-016-0075-5. eCollection 2016. PMID 27252778
- [Background] Sijbrandij M, Farooq S, Bryant RA, Dawson K, Hamdani SU, Chiumento A, Minhas F, Saeed K, Rahman A, van Ommeren M. Problem Management Plus (PM+) for common mental disorders in a humanitarian setting in Pakistan; study protocol for a randomised controlled trial (RCT). BMC Psychiatry. 2015 Oct 1;15:232. doi: 10.1186/s12888-015-0602-y. PMID 26428314
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Derived] Sangraula M, Van't Hof E, Luitel NP, Turner EL, Marahatta K, Nakao JH, van Ommeren M, Jordans MJD, Kohrt BA. Protocol for a feasibility study of group-based focused psychosocial support to improve the psychosocial well-being and functioning of adults affected by humanitarian crises in Nepal: Group Problem Management Plus (PM+). Pilot Feasibility Stud. 2018 Jul 18;4:126. doi: 10.1186/s40814-018-0315-3. eCollection 2018. PMID 30038793